CLINICAL TRIAL: NCT07219719
Title: Temporal Interference for Thalamocortical Activity and Network Modulation
Acronym: TITAN
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-1275; SMPH/PSYCHIATRY/PSYCHIATRY (Other: UW Madison); Protocol Version 10/20/25 (Other: UW Madison)
Record Dates: First submitted 2025-10-16; First posted 2025-10-22 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants

STUDY DESIGN:
Intervention Model Description: This pilot study employs a within-subject, counterbalanced crossover design in which each participant serves as their own control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Stimulation (Experimental): Participants will complete two stimulation phases-overnight TI-TES during non-rapid eye movement (NREM) sleep and TI-TES during quiet wakefulness
  Interventions: Device: Temporal Interference Transcranial electrical stimulation (TI-TES)

INTERVENTIONS:
Device: Temporal Interference Transcranial electrical stimulation (TI-TES) — TI-TES uses specific electrode arrangement patterns to selectively stimulate the brain. Participants will wear an hdEEG (high density electroencephalography) cap which will allow intermittent periods of stimulation from TI-TES.

SUMMARY:
The goal of this clinical trial is to find out whether a type of electrical brain stimulation, called temporal interference stimulation, can temporarily change the way different parts of the brain communicate with each other.

Participants will:

* Complete two stimulation phases - overnight and during wakefulness
* Undergo two MRIs per study phase

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of personalized thalamic temporal interference transcranial electrical stimulation (TI-TES) to modulate thalamocortical activity and connectivity in healthy adults. Using a within-subject, counterbalanced crossover design, participants will complete two stimulation phases: (1) repeated overnight TI-TES during NREM sleep and (2) repeated TI-TES during quiet wakefulness. Each phase consists of two sessions. Phases are separated by a ≥4-week washout. Resting-state functional magnetic resonance imaging (fMRI) will be acquired before and after each phase to assess sustained changes in thalamocortical functional connectivity, with high-density EEG providing secondary measures of brain-state-specific oscillatory modulation (sigma/spindles in sleep, alpha in wake).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-50
* Medically healthy
* U.S. citizen or holding permanent resident status
* English-speaking

Exclusion Criteria:

* Any current or past history of neurological disorders or acquired neurological disease (e.g. stroke, traumatic brain injury), including intracranial lesions (including clinically significant findings identified in first MRI)
* History of inpatient psychiatric hospitalization
* History of head trauma resulting in prolonged loss of consciousness; or a history of greater than 3 grade I concussions
* Current history of poorly controlled headaches including intractable or poorly controlled migraines
* Any systemic illness or unstable medical condition that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
* History of seizures, diagnosis of epilepsy, history of abnormal (epileptiform) EEG, or family history of treatment resistant epilepsy except for a single seizure of benign etiology (e.g. febrile seizures) in the judgment of a board-certified neurologist
* Possible pregnancy or plan to become pregnant in the next 6 months (self reported)
* Any metal in the head
* Any medical devices or implants (i.e. cardiac pacemaker, medication infusion pump, cochlear implant, vagal nerve stimulator)
* Dental implants
* Permanent retainers
* Any hair braid, dreadlocks, hair pieces, or extensions which cannot be taken out before the study sessions
* Any head coverings or headdress that participant feels uncomfortable removing for the purposes of study sessions
* Any medication that may alter seizure threshold taken during the study i.e., Attention-deficit/hyperactivity disorder (ADHD) stimulants (Adderall, amphetamine); Tricyclic/atypical antidepressants (amitriptyline, doxepin, imipramine, maprotiline, nortriptyline, bupropion); Antipsychotics (chlorpromazine, clozapine), Bronchodilators (theophylline, aminophylline); Antibiotics (fluoroquinolones, imipenem, penicillin, cephalosporins, metronidazole, isoniazid); Antivirals (valacyclovir, ritonavir); over the counter antihistamines (diphenhydramine, Benadryl)
* Claustrophobia (a fear of small or closed places)
* Back problems that would prevent lying flat for up to two hours
* Regular night-shift work (second or third shift)
* Sleep apnea or other sleep disorder (self-reported)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in thalamocortical functional connectivity (FC): resting state fMRI | Pre- to post-intervention, up to 2 weeks
  Resting-state fMRI will be used to assess changes in thalamocortical functional connectivity before and after repeated thalamic TI-TES delivered during NREM sleep and quiet wakefulness.
Difference in magnitude of FC changes between sleep and wake | 8 weeks
  The magnitude of FC changes between sleep and wake stimulation phases will be evaluated.
Difference in spatial distribution of FC changes between sleep and wake | 8 weeks
  The spatial distribution of FC changes between sleep and wake stimulation phases will be evaluated.

SECONDARY OUTCOMES:
Change in sigma-band power (EEG, sleep phase) | During and after each overnight stimulation session, up to 1 week
  Sigma band power will be measured with high density EEG (hdEEG) during stimulation, and will be analyzed to quantify stimulation-related changes in sigma-band power during NREM sleep.
Change in alpha band power during wake stimulation sessions | During and after each wake stimulation session, up to 1 week
  Alpha band power will be measured with hdEEG during stimulation, and will be analyzed to quantify stimulation-related changes in alpha-band power during quiet wakefulness stimulation.
Return to baseline thalamocortical FC | 8 weeks
  After the ≥4-week washout, thalamocortical FC will be assessed by resting-state fMRI prior to the second stimulation phase.
Change in structural thalamocortical connectivity | Pre- to post-intervention, up to 2 weeks
  Will be measured using diffusion-weighted imaging (DWI) in each phase.
Change in mood | Baseline to 12 weeks
  Mood will be scored using Positive and Negative Affect Schedule (PANAS). PANAS is a 20 item questionnaire, each item is rated on a 5-point scale, with 1 = "Very slightly or not at all" and 5 = "Extremely". To score PANAS, sum the scores for the 10 Positive Affect (PA) items and the 10 Negative Affect (NA) items separately on the 5-point scale. Higher scores for PA indicate a greater degree of positive emotion, while higher scores for NA indicate more negative emotion, with both scales ranging from 10 (low affect) to 50 (high affect).
Change in Boston Cognitive Assessment (BoCA) | Baseline to 12 weeks
  BoCA™ evaluates eight cognitive domains using randomized, non-repeating tasks to minimize practice effects. The total maximum score is 30. Higher scores indicate better cognitive performance.
Change in spindle characteristics: Density | Up to 1 week
  HdEEG will be analyzed to assess stimulation-related changes in spindle density during NREM sleep.
Change in spindle characteristics: Amplitude | Up to 1 week
  HdEEG will be analyzed to assess stimulation-related changes in spindle amplitude during NREM sleep.
Change in spindle characteristics: Duration | Up to 1 week
  HdEEG will be analyzed to assess stimulation-related changes in spindle duration during NREM sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Albantakis, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes